CLINICAL TRIAL: NCT03102190
Title: Phase Ib/II Clinical Trial of Topical Verapamil Hydrochloride for Chronic Rhinosinusitis With Nasal Polyps
Brief Title: Trial of Topical Verapamil in Chronic Rhinosinusitis With Nasal Polyps
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Phase II funding not available
Sponsor: Benjamin Bleier (Other)
Responsible Party: Sponsor-Investigator, Benjamin Bleier, Principal Investigator, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17-002H
Record Dates: First submitted 2017-02-14; First posted 2017-04-05 (Actual); Results first posted 2019-06-21 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Sinusitis; Nasal Polyps
MeSH Terms: conditions — Sinusitis; Nasal Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase Ib (Experimental): The phase Ib study will consist of an accelerated titration, intrapatient dose escalation cohort, with double-dose step design of Verapamil Hydrochloride. Intranasal BID for 1 week. Dose escalation will occur weekly as a doubling of the dose from 10-120mg Verapamil delivered in 240mL buffered normal saline. If a single, any course, dose-limiting toxicity (DLT) or second, any course, IT occurs, two additional patients will be recruited at that identified dose and Phase Ib will revert to a standard 3+3 design. If any patient un-enrolls while the dose escalation is still occurring, they will be replaced to maintain 3 patient cohorts. The maximal administered dose (MAD) will be considered that at which at least 2 DLTs or 4 ITs occur and the MTD will then be assigned to the immediate preceding dose.
  Interventions: Drug: Verapamil Hydrochloride Intranasal

INTERVENTIONS:
Drug: Verapamil Hydrochloride Intranasal — Verapamil solution for injection, supplied in vials, will be utilized in a Neil Med Sinus Rinse of 240mL buffered normal saline.

SUMMARY:
Verapamil is an L-type calcium channel blocker(CCB) which has been shown to reduce inflammation in a variety of tissues. Chronic rhinosinusitis with nasal polyps (CRSwNP) is characterized by eosinophilic inflammation as well as P-gp overexpression. A previous trial of oral Verapamil showed preliminary efficacy for the treatment of CRSwNP. The goal of this study is to evaluate the safety and efficacy of intranasal Verapamil in CRSwNP. The study was initially approved as a Phase Ib/II, but only the Phase Ib portion was completed as part of this protocol.

DETAILED DESCRIPTION:
CRSwNP is a prevalent disease associated with major direct and indirect costs. Acute and Chronic Rhinosinusitis are estimated to affect up to 16% of the US population. They account for approximately 11 million or 1% of all office visits per year in the US and are the most common cause for antibiotic prescriptions in the community. CRS alone impacts more than 30 million Americans resulting in $6.9 to $9.9 billion in annual healthcare expenditures and $12.8 billion in productivity costs. The subset of patients in Europe with CRSwNP has been estimated to be between 2 and 4.3% and is thought to be similar in the US. This population remains one of the most challenging subgroups of CRS to manage effectively.

Recent evidence has focused on the sinonasal epithelial cell as a primary driver of the local dysregulated immune response through secretion of type 2 helper T-cell(Th2) promoting cytokines. While these studies suggest that epithelial cells are capable of orchestrating a local immune response, the mechanisms responsible for regulating cytokine secretion are poorly understood and may be influenced by the efflux function of epithelial P-glycoprotein(P-gp). Studies by the investigator's group have demonstrated that P-gp is overexpressed in the mucosa of patients with Th2 skewed CRS endotypes including CRSwNP and is capable of regulating the secretion of Th2 polarizing cytokines. Together, these findings suggest that P-gp participates in the non-canonical regulation of cytokine secretion within CRSwNP and may thereby represent a druggable target.

The investigator's group therefore undertook a randomized, double-blind, placebo-controlled trial to test the efficacy of low dose oral Verapamil HCl, a known first generation P-gp inhibitor, for the treatment of CRSwNP. Our findings demonstrated significant efficacy in both of the primary and secondary endpoints with no significant side effects. However, a logistic regression analysis revealed two important relationships between baseline characteristics and efficacy. First, patients with elevated BMI had significantly lower improvements in the Sinonasal Outcome Test (SNOT-22) (p=0.01). The second is that patients with the highest total mucus P-gp levels experienced less benefit(p=0.01).

While Verapamil HCl has significant potential for the treatment of CRSwNP through P-gp inhibition, higher doses must be achieved to extend the effect to patients with elevated BMIs and the highest levels of P-gp expression. As increasing oral dosing could result in cardiac side effects, topical delivery represents a promising alternative. As exosome bound P-gp may be more stable and representative of disease state than total mucus P-gp concentration, exosomal P-gp demands further exploration as a novel biomarker of disease severity and drug response.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the Mass Eye and Ear Sinus Center
* Age 18-80 yrs old
* Diagnosed with Chronic Rhinosinusitis with Nasal Polyps according to the EPOS 2012 consensus criteria
* Post-operative with a Lund-Kennedy Poly score of <4
* Baseline SNOT-22 Score ≥ 30

Exclusion Criteria:

* Patients with the following comorbidities:
* GI Hypomotility
* Heart Failure
* Liver Failure
* Kidney Disease
* Muscular Dystrophy
* Pregnant or Nursing Females
* Steroid Dependency
* Hypertrophic Cardiomyopathy
* Any Atrial or Ventricular arrhythmia (ie. Atrial fibrillation, atrial flutter, etc..)
* Resting Heart Rate less than 60 beats per minute
* Baseline Systolic Blood Pressure less than 110 mmHg
* Baseline Diastolic Blood Pressure less than 70 mmHg
* Baseline Mean Arterial Pressure Less than 60 mmHg
* PR interval less than 0.12 seconds
* Patients taking the following medications:
* Aspirin
* Beta-blockers
* Cimetidine(Tagamet)
* Clarithromycin(Biaxin)
* Cyclosporin
* Digoxin
* Disopyramide(Norpace)
* Diuretics
* Erythromycin
* Flecainide
* HIV Protease Inhibitors(Indinavir, Nelfinavir, Ritonavir)
* Quinidine
* Lithium
* Pioglitazone
* Rifampin
* St Johns Wort
* Patients with cardiac or conduction abnormality picked up by screening EKG
* Post-op patients with surgery within 3 months prior to enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin S Bleier, MD, Principal Investigator — Massachusetts Eye and Ear
Locations (1):
- Massachusetts Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miyake MM, Nocera A, Levesque P, Guo R, Finn CA, Goldfarb J, Gray S, Holbrook E, Busaba N, Dolci JEL, Bleier BS. Double-blind placebo-controlled randomized clinical trial of verapamil for chronic rhinosinusitis with nasal polyps. J Allergy Clin Immunol. 2017 Jul;140(1):271-273. doi: 10.1016/j.jaci.2016.11.014. Epub 2017 Jan 23. No abstract available. PMID 28126245
- [Background] Meltzer EO, Hadley J, Blaiss M, Benninger M, Kimel M, Kleinman L, Dupclay L, Garcia J, Leahy M, Georges G. Development of questionnaires to measure patient preferences for intranasal corticosteroids in patients with allergic rhinitis. Otolaryngol Head Neck Surg. 2005 Feb;132(2):197-207. doi: 10.1016/j.otohns.2004.10.010. PMID 15692526
- [Background] Chin D, Harvey RJ. Nasal polyposis: an inflammatory condition requiring effective anti-inflammatory treatment. Curr Opin Otolaryngol Head Neck Surg. 2013 Feb;21(1):23-30. doi: 10.1097/MOO.0b013e32835bc3f9. PMID 23172039
- [Background] Poetker DM, Jakubowski LA, Lal D, Hwang PH, Wright ED, Smith TL. Oral corticosteroids in the management of adult chronic rhinosinusitis with and without nasal polyps: an evidence-based review with recommendations. Int Forum Allergy Rhinol. 2013 Feb;3(2):104-20. doi: 10.1002/alr.21072. Epub 2012 Aug 7. PMID 22887970
- [Background] Khakzad MR, Mirsadraee M, Mohammadpour A, Ghafarzadegan K, Hadi R, Saghari M, Meshkat M. Effect of verapamil on bronchial goblet cells of asthma: an experimental study on sensitized animals. Pulm Pharmacol Ther. 2012 Apr;25(2):163-8. doi: 10.1016/j.pupt.2011.11.001. Epub 2011 Nov 25. PMID 22133887
- [Background] Matsumori A, Nishio R, Nose Y. Calcium channel blockers differentially modulate cytokine production by peripheral blood mononuclear cells. Circ J. 2010 Mar;74(3):567-71. doi: 10.1253/circj.cj-09-0467. Epub 2010 Jan 30. PMID 20118567
- [Background] Li G, Qi XP, Wu XY, Liu FK, Xu Z, Chen C, Yang XD, Sun Z, Li JS. Verapamil modulates LPS-induced cytokine production via inhibition of NF-kappa B activation in the liver. Inflamm Res. 2006 Mar;55(3):108-13. doi: 10.1007/s00011-005-0060-y. PMID 16673153
- [Background] Becker WJ. Cluster headache: conventional pharmacological management. Headache. 2013 Jul-Aug;53(7):1191-6. doi: 10.1111/head.12145. Epub 2013 Jun 14. PMID 23773141
- [Background] Lanteri-Minet M, Silhol F, Piano V, Donnet A. Cardiac safety in cluster headache patients using the very high dose of verapamil (>/=720 mg/day). J Headache Pain. 2011 Apr;12(2):173-6. doi: 10.1007/s10194-010-0289-x. Epub 2011 Jan 22. PMID 21258839
- [Background] Hopkins C, Gillett S, Slack R, Lund VJ, Browne JP. Psychometric validity of the 22-item Sinonasal Outcome Test. Clin Otolaryngol. 2009 Oct;34(5):447-54. doi: 10.1111/j.1749-4486.2009.01995.x. PMID 19793277
- [Background] Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, Cohen N, Cervin A, Douglas R, Gevaert P, Georgalas C, Goossens H, Harvey R, Hellings P, Hopkins C, Jones N, Joos G, Kalogjera L, Kern B, Kowalski M, Price D, Riechelmann H, Schlosser R, Senior B, Thomas M, Toskala E, Voegels R, Wang de Y, Wormald PJ. European Position Paper on Rhinosinusitis and Nasal Polyps 2012. Rhinol Suppl. 2012 Mar;23:3 p preceding table of contents, 1-298. PMID 22764607
- [Background] Klossek JM, Neukirch F, Pribil C, Jankowski R, Serrano E, Chanal I, El Hasnaoui A. Prevalence of nasal polyposis in France: a cross-sectional, case-control study. Allergy. 2005 Feb;60(2):233-7. doi: 10.1111/j.1398-9995.2005.00688.x. PMID 15647046

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase Ib
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Phase Ib
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity
Description: Dose Limiting Toxicity will be defined as a development of 2nd or 3rd degree heart block as measured by an EKG. (Phase Ib primary outcome)
Time Frame: 1-8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib
Number analyzed (Participants) | 6
Participants | 0
Statistical Analysis 1: Comparison: Phase Ib; Test type: Other; The analysis of the safety endpoints will be presented with means and standard deviations of their occurrence within the study population. The safety of the drug will be determined by analyzing the rate of adverse events in both phases of the trial. An occurrence of 10% within the study population will be considered significant

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Phase Ib
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase Ib (N=6)
Low heart rate (Cardiac disorders) | 1 (3)
Headache (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT03102190/Prot_SAP_000.pdf